CLINICAL TRIAL: NCT00928174
Title: Measurement of Anti-Androgen Response Using Fluorine-18 Fluorocholine PET/CT in Androgen-Insensitive Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Queen's Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sandi Kwee, Sandi A. Kwee, M.D., Queen's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RA-2009-009; R21CA139687 (NIH)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: Androgen insensitive prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Fluorine-18 fluorocholine IV in conjunction with PET/CT imaging, up to 3 doses.
  Interventions: Drug: IV administration of fluorine-18 fluorocholine followed by PET/CT imaging

INTERVENTIONS:
Drug: IV administration of fluorine-18 fluorocholine followed by PET/CT imaging — Imaging intervention performed prior to and 30-75 days post a change in anti-androgen therapy.

SUMMARY:
The purpose of this study is to determine whether positron emission tomography / computed tomography (PET/CT) using fluorine-18 fluorocholine as an imaging agent can characterize regional responses to anti-androgen therapies in a manner that in the future aid in the customized planning of treatments for patients with androgen-insensitive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Men, over 18 years of age, with histologically-confirmed diagnosis of prostate cancer
3. History of treatment by complete androgen blockade for greater than 3 months prior to enrollment
4. Serum testosterone level < 50 ng/ml. Castrate testosterone levels must be from orchiectomy or current therapy with leutinizing hormone-releasing hormone agonist.
5. Progressive disease evidenced by two consecutive rises in prostate specific antigen (PSA) above a nadir value, with the absolute value of the latest PSA > 2. 0 ng/ml.
6. Patient will be undergoing a therapeutic intervention under the supervision of his treating physician (urologist, oncologist).

Exclusion Criteria:

1. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or superficial transitional cell carcinoma of the bladder.
2. Serious underlying medical conditions that would otherwise impair the patient's ability to undergo imaging.
3. Patient weighs over 350 lbs (due to scanner weight limit).
4. Clinical life expectancy < 12 weeks.
5. Participated in other radioactive drug studies where estimated total cumulative dose within 1 year is > 0.05 Sievert for whole body, active blood-forming organs, eye lens, gonads, or 0.15 Sievert for other organs.
6. Concurrent Therapy. Allowed: prior hormonal therapy; concurrent leuteinizing hormone releasing hormone (LHRH) agonist; prior surgery; prior or concurrent bisphosphonate. Not allowed: concurrent anti-androgen or secondary hormonal therapy, prior or concurrent chemotherapy, concurrent radiotherapy or radioisotope therapy (e.g., strontium). Other: Prior radiotherapy or radioisotope therapy must be > 12 weeks since last treatment.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandi A Kwee, MD, Principal Investigator — The Queen's Medical Center
Locations (1):
- The Queen's Medical Center, Honolulu, Hawaii, United States

REFERENCES:
- [Derived] Lee J, Sato MM, Coel MN, Lee KH, Kwee SA. Prediction of PSA Progression in Castration-Resistant Prostate Cancer Based on Treatment-Associated Change in Tumor Burden Quantified by 18F-Fluorocholine PET/CT. J Nucl Med. 2016 Jul;57(7):1058-64. doi: 10.2967/jnumed.115.169177. Epub 2016 Feb 16. PMID 26912444

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Fluorine-18 fluorocholine IV in conjunction with PET/CT imaging, up to 3 doses.
  IV administration of fluorine-18 methylcholine followed by PET/CT imaging: Imaging intervention performed prior to and 30-75 days post a change in anti-androgen therapy.
Period: Overall Study
Arm/Group | Single Arm
Started | 27
Completed | 22 (3 withdrawn before start of participation)
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 27
Age, Customized [Number; unit: participants] — Age (10-year groupings)
  participants
    <40 | 0
    40-49 years | 0
    50-59 years | 1
    60-69 years | 9
    70-79 years | 4
    80-89 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Outcome Correspondence to Imaging Results With Fluorine-18 Fluorocholine PET/CT
Description: The percentage of patients within a given prostate specific antigen range found to have at least one abnormal lesion demonstrating increased fluorine-18 fluorocholine uptake on positron emission tomography (PET) imaging consistent with the clinical diagnosis of metastatic or recurrent prostate cancer.
Time Frame: Concurrent with PET Procedure
Population: Outcome Measure Data Table reflects data from the 22 subjects completing the current study.
Measure: Number; unit: %PET-positive cases in a given PSA range
Groups:
- Single Arm: fluourine-18 fluorocholine IV in conjunction with PET/CT imaging, up to 3 doses.
  IV administration of fluorine-18 fluoromethylcholine followed by PET/CT imaging: Imaging intervention performed prior to and 30-75 days post a change in anti-androgen therapy.
Arm/Group | Single Arm
Number analyzed (Participants) | 22
%PET-positive cases in a given PSA range
  PSA > 4 ng/mL (19 cases) | 100
  PSA 2-4 ng/mL (2 cases) | 100
  PSA > 0.5 - 2 ng/mL (1 cases) | 100
  PSA <= 0.5 ng/mL (0 cases) | 0

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes